CLINICAL TRIAL: NCT00468390
Title: Capsaicin-Evoked Pain in Patients With Complex Regional Pain Syndrome
Brief Title: Capsaicin-Evoked Pain in Patients With CRPS
Status: Completed | Type: Observational
Sponsor: Danish Pain Research Center (Other)
Other Study IDs: Capsaicin in CRPS
Record Dates: First submitted 2007-05-01; First posted 2007-05-02 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: CRPS (Complex Regional Pain Syndromes)
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the effect of capsaicin in patients with Complex Regional Pain Syndrome.

DETAILED DESCRIPTION:
Primary outcome parameters: Capsaicin-induced pain and inflammation.

Secondary outcome parameters: Peripheral sensory and autonomic function.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 or older.
* Pain in arm or hand > 3 months.
* Diagnosed with CRPS acc. to diagnostic research criteria (Harder et al., 2005)
* Inclusion of healthy subjects: age-, gender-, and BMI-matched.

Exclusion Criteria:

* Other significant disease affecting the parameters measured, including cardiovascular disease.
* Treatment with anticholinergics, sympathomimetics and parasympathomimetics, and alpha- and beta-adrenergics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2007-04; Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Troels S Jensen, MD, DMSc, Study Chair — Danish Pain Research Center, Aarhus University Hospital
Locations (1):
- Danish Pain Research Center, Aarhus University Hospital, Aarhus, Denmark